CLINICAL TRIAL: NCT05333965
Title: To Evaluate The Performance Of Two Monthly Replacement Silicone Hydrogel Contact Lenses After 1-month Of Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-132
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A, Then Lens B (Experimental): Participants wore Lens A for one month and then crossed over to wear Lens B for one month.
  Interventions: Device: Lens A (lehfilcon A lens); Device: Lens B (comfilcon A lens)
- Lens B, Then Lens A (Experimental): Participants wore Lens B for one month and then crossed over to wear Lens A for one month.
  Interventions: Device: Lens A (lehfilcon A lens); Device: Lens B (comfilcon A lens)

INTERVENTIONS:
Device: Lens A (lehfilcon A lens) — Daily wear for 1 month.
Device: Lens B (comfilcon A lens) — Daily wear for 1 month.

SUMMARY:
To evaluate the performance of two monthly replacement silicone hydrogel contact lenses in habitual FRP CL wearers when worn for 1-month.

DETAILED DESCRIPTION:
This study will be a prospective, randomized, double-masked, single-site, 1-month cross-over design involving bilateral eye daily wear of two different monthly replacement CL types. Each lens will be worn bilaterally for approximately one month.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 17 years of age and has full legal capacity to volunteer;
2. Self-reports having had a full eye examination within the previous 2 years;
3. Has read and signed an information consent letter;
4. Is willing and able to follow instructions and maintain the appointment schedule;
5. Is a habitual wearer of frequent replacement contact lenses;
6. Anticipates no difficulty wearing the contact lenses for 6 days/week and 8 hours/day during the study;
7. Has refractive astigmatism no higher than -0.75DC in each eye;
8. Can be successfully fit with both study lens types;
9. Achieves at least 0.4 logMAR VA monocularly and at least 0.2 logMAR VA binocularly with each study lens type.

Exclusion Criteria:

1. Is participating in any concurrent clinical research study;
2. Has any known active ocular disease and/or infection;
3. Has an unstable systemic condition that in the opinion of the investigator may affect vision or contact lens comfort across the 2-month study duration;
4. Is using any systemic or topical medications in an irregular routine that in the opinion of the investigator may affect vision or contact lens comfort across the 2-month study duration;
5. Has known sensitivity to the diagnostic sodium fluorescein to be used in the study;
6. Is an employee of the Centre for Ocular Research & Education.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD FCOptom, Principal Investigator — Centre for Ocular Research and Education
Locations (1):
- School of Optometry & Vision Science, Waterloo, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 27 people screened and 26 were dispensed with study products. Two participants discontinued and 24 completed the study.
Groups:
- Lens A, Then Lens B: Participants wore Lens A for one month and then crossed over to wear Lens B for one month. Each Lens type was worn on a daily wear basis for one month.
- Lens B, Then Lens A: Participants wore Lens B for one month and then crossed over to wear Lens A for one month. Each Lens type was worn on a daily wear basis for one month.
Period: First Intervention
Arm/Group | Lens A, Then Lens B | Lens B, Then Lens A
Started | 13 | 13
Completed | 13 | 11
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Lens A, Then Lens B | Lens B, Then Lens A
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Analysis Population: Out of 26 participants, 2 of them discontinued. Therefore, overall base participants (Analysis population) are 24.
Arm/Group | Analysis Population
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lens Handling on Lens Removal
Description: Lens handling on removal will be measured on a scale of 0-10, 0.5 steps (0=Completely dissatisfied,10=Completely satisfied)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lens A: Participants wore Lens A for 1 month.
- Lens B: Participants wore Lens B for 1 month.
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 24 | 24
units on a scale | 8.4 (2.3) | 8.9 (1.3)

ADVERSE EVENTS:
Time Frame: From dispense up to one month on each study lens, for total of two months
Description: Enrollment population (n=26)
Arm/Group | Lens A | Lens B
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 1/26
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lens A (N=26) | Lens B (N=26)
Significant Ocular Redness (Eye disorders) | 0 (0) | 1 (2)
asymptomatic corneal infiltrate keratitis (Eye disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT05333965/Prot_SAP_000.pdf